CLINICAL TRIAL: NCT03722134
Title: Mechanochemical Ablation vs Thermal Ablation in Patients With Great Saphenous Vein Insufficiency
Brief Title: Mechanochemical Ablation vs Thermal Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Maarit Venermo, Professor of Vascular Surgery, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Clarivein RCT
Record Dates: First submitted 2018-10-23; First posted 2018-10-26 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2018-10

CONDITIONS: Varicose Veins of Lower Limb
Keywords: Great saphenous vein; Thermal ablation; Mechanochemical ablation; Randomized controlled trial

STUDY DESIGN:
Intervention Model Description: Our study aim was to assess the applicability and safety of MOCA in short term as well as occlusion rate and disease specific quality of life one year after the procedure, and compare it with currently used thermal ablation methods of laser ablation (EVLA) and radiofrequency ablation (RFA) in a randomized controlled trial.
  Randomization took place by a study nurse after the appointment, using block randomization with sealed envelopes into EVLA, RFA, or MOCA in ratio 1:1:2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- MOCA (Experimental): The refluxing GSV was treated with ClariVein catheter (endovenous mechanochemical ablation).
  Interventions: Procedure: MOCA
- EVLA (Active Comparator): The refluxing GSV was treated with endovenous laser ablation.
  Interventions: Procedure: EVLA
- RFA (Active Comparator): The refluxing GSV was treated with radiofrequency ablation.
  Interventions: Procedure: RFA

INTERVENTIONS:
Procedure: MOCA — Great saphenous vein occlusion with a mechanochemical chateter which cause mechanical injury to vessel intima and gives sclerosant to the intima.
  Arms: MOCA
Procedure: EVLA — Great saphenous vein occlusion with a thermal laser chateter
  Arms: EVLA
Procedure: RFA — Great saphenous vein occlusion with a thermal radiofrequency chateter
  Arms: RFA

SUMMARY:
Patients with GSV reflux were randomized to undergo either MOCA or thermal ablation with laser or radiofrequency. The main outcome measure was the occlusion rate of the GSV at one year.Patients with GSV reflux were randomized to undergo either MOCA or thermal ablation with laser or radiofrequency. The main outcome measure was the occlusion rate of the GSV at one and three years.

DETAILED DESCRIPTION:
During 2014-2015, all patients referred to our vascular surgery clinic by their general practitioners due to varicose veins were screened for GSV insufficiency. We invited all patients filling the inclusion criteria to participate in this study.

Included patients were randomized to receive either thermal ablation (laser ablation or radiofrequency ablation) or mechanochemical ablation with the Clarivein device to treat the refluxing GSV.

The patients filled the Aberdeen Varicose Veins Questionnaire (AVVQ) at the baseline. We recorded the preoperative diameter of the GSV, specifically the diameter at the most proximal 20 centimetres, and the mean overall diameter at the thigh.

During the procedure, before discharge, and a week after, the patients reported pain scores using Visual Analogue Scale (VAS) on a scale of 0 to 10. At the one-month follow-up visit, we recorded wound healing, haematomas or bruising, nerve injuries, and pigmentation. The status of the GSV was examined with duplex Doppler ultrasound. The patients were also asked to determine what would have been the optimal sick leave after the procedure.

At the one-year follow-up, nerve injuries, pigmentation, and clinical status were recorded, as well as the status of the GSV with duplex Doppler ultrasound. The patients also filled the AVVQ questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* clinical classification of venous disease C2-C4
* ultrasound-verified reflux in the GSV
* mean GSV diameter in the thigh between 5 and 12 millimetres
* informed consent.

Exclusion Criteria:

* body mass index (BMI) of over 40
* peripheral arterial disease
* lymphoedema
* pregnancy
* allergy to either the sclerosant or lidocaine
* severe general illness
* malignancy
* previous deep venous thrombosis
* previous varicose vein intervention in the same leg
* coagulation disorders

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Occlusion rate | One year after the treatment
  Occlusion rate of the great saphenous vein
Freedom from reflux | One year after the treatment
  The absence of reflux in the treated great saphenous vein
Disease-specific quality of life | One year after the treatment
  Quality of life as measured by the Aberdeen Varicose Veins Questionnaire
Occlusion rate | three years after the treatment
  Occlusion rate of the great saphenous vein
Freedom from reflux | three years after the treatment
  The absence of reflux in the treated great saphenous vein
Disease-specific quality of life | three years after the treatment
  Quality of life as measured by the Aberdeen Varicose Veins Questionnaire
Occlusion rate | five years after the treatment
  Occlusion rate of the great saphenous vein
Freedom from reflux | five years after the treatment
  The absence of reflux in the treated great saphenous vein
Disease-specific quality of life | five years after the treatment
  Quality of life as measured by the Aberdeen Varicose Veins Questionnaire

SECONDARY OUTCOMES:
Peroperative and immediate postoperative pain | During the procedure, immediately after, and at one week after the treatment
  Perceived pain using Visual Analogue Scale (Range 0-10; 0=no pain; 2=Mild pain, 4=Nagging, uncomfortable pain; 6= Miserable pain; 8=Horrible pain; 10=worst possible, unbearable pain)
Sick leave | During the immediate postoperative period up to one month
  Number of sick leave days necessary after the treatment
Pain medication | During the immediate postoperative period up to one month
  The amount and type of pain medication received during and after the treatment
30-day occlusion rate | 30 days after the treatment
  The occlusion rate of the treated great saphenous vein
Complications | Up to five years after the treatment
  All complications (deep venous thrombosis, nerve injuries, infections etc) after the treatment

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vahaaho S, Halmesmaki K, Mahmoud O, Alback A, Noronen K, Venermo M. Three-year results of a randomized controlled trial comparing mechanochemical and thermal ablation in the treatment of insufficient great saphenous veins. J Vasc Surg Venous Lymphat Disord. 2021 May;9(3):652-659. doi: 10.1016/j.jvsv.2020.08.007. Epub 2020 Aug 12. PMID 32795619
- [Derived] Vahaaho S, Mahmoud O, Halmesmaki K, Alback A, Noronen K, Vikatmaa P, Aho P, Venermo M. Randomized clinical trial of mechanochemical and endovenous thermal ablation of great saphenous varicose veins. Br J Surg. 2019 Apr;106(5):548-554. doi: 10.1002/bjs.11158. PMID 30908611